CLINICAL TRIAL: NCT04414293
Title: Phase II Study of Low Dose Pulmonary Irradiation in Patients With COVID-19 Infection of Bad Prognosis
Brief Title: Low Dose Pulmonary Irradiation in Patients With COVID-19 Infection of Bad Prognosis
Acronym: COVRTE-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Provincial de Castellon (Other)
Responsible Party: Principal Investigator, Carlos Ferrer Albiach, MD, Hospital Provincial de Castellon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FHPCS-20-001
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: COVID; Pneumonia, Viral
Keywords: covid-19 pneumonia; Low dose Radiotherapy
MeSH Terms: conditions — Pneumonia, Viral | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): All the patients will be treated with low dose lung radiation
  Interventions: Radiation: Lung Low Dose Radiation

INTERVENTIONS:
Radiation: Lung Low Dose Radiation — The administration of low-dose lung radiation produces anti-inflammatory effects that will decrease the pulmonary inflammatory response.

SUMMARY:
The administration of low-dose lung irradiation produces anti-inflammatory effects that will decrease the pulmonary inflammatory response.

The present study will evaluate the efficacy of treatment with low-dose pulmonary radiotherapy added to standard support therapy, in hospitalized patients with respiratory symptoms due to COVID-19 pneumonia, who do not experience improvement with conventional medical therapy and are not subsidiaries of ICU

DETAILED DESCRIPTION:
The WHO has officially confirmed that: "Currently, there is no specific pharmacological available treatment for COVID-19".

Beyond vital support, there are not currently treatment options for Coronavirus disease (COVID-19) and related pneumonia, the infection caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Pulmonary irradiation is an option for the treatment of COVID-19 pneumonia and could be available quickly and with a duration of about 15 minutes of treatment.

Thoracic irradiation therapy at very low doses (0.5-1.0 Gy) dates back to the 1920s and was the only effective mean to treat certain infectious and inflammatory diseases prior to the development of antimicrobial therapies in the 1940s.

The goal is to replicate low-dose radiation therapy, just as it was used 80 years ago for viral pneumonia with great success. It will be administered for a new disease, pneumonia caused by COVID-19, for which there is no cure and many people are dying, mainly from severe acute respiratory syndrome leading to very severe hypoxemic acute respiratory failure refractory to treatment.

This therapy is expected to remedy acute respiratory syndrome by reducing inflammation, and it also has a low risk of side effects and toxicities, given the low doses received, more than one hundred times lower, compared to the usual radiotherapy used to tumor treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years old
* Hospitalized with COVID-19 positive not subsidiary of ICU with severe disease defined by the presence of ALL the following characteristics:

  * Presence of unilateral or bilateral pulmonary infiltrates in chest X-ray or computed tomography (CT).
  * Acute respiratory failure expressed by PaO2 / FIO2 <300.
  * Lymphopenia ≤0.8 × 109 / L (800 lymphocytes / ml).
  * Patients with ≤8 days from the onset of symptoms.

Exclusion Criteria:

* Patient not consent to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
blood oxygen saturation level | 48 hours
  Clinical improvement of respiratory symptoms due to COVID-19 pneumonia after the treatment, measured as blood oxygen saturation levels
Torax X-ray | 48 hours
  radiological improvement of respiratory symptoms due to COVID-19 pneumonia after the treatment.

SECONDARY OUTCOMES:
Hospitalization | 2 months
  number of days of hospital stay.
days free of assisted mechanical respiration | 3 month
  Number of days free of assisted mechanical respiration.
Mortality | 3 months
  number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ferrer Albiach, MD, Principal Investigator — Hospital Provincial de Castellon
Locations (1):
- Hospital Provincial de Castellon, Castellon, Castellon, Spain